CLINICAL TRIAL: NCT03719352
Title: Analysis, Comparison and Evaluation of Cervical Range of Motion and Neck Pain After Deep Dry Needling and Superficial Dry Needling in the Upper Trapezius: A Randomised Controlled Trial
Brief Title: Superficial Dry Needling Versus Deep Dry Needling on the Upper Trapezius
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, SERGIO MONTERO NAVARRO, Principal Investigator, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEU UCH 205
Record Dates: First submitted 2018-10-15; First posted 2018-10-25 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (participant, outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Deep dry needling (Experimental): Deep dry needling will be applied in the upper trapezius myofascial trigger point
  Interventions: Procedure: Experimental: Deep dry needling
- Superficial dry needling (Experimental): Superficial dry needling will be applied in the upper trapezius myofascial trigger point
  Interventions: Procedure: Experimental: Superficial dry needling
- Placebo Gastrocnemius dry needling (Placebo Comparator): A technique simulating dry needling will be applied in the gastrocnemius myofascial trigger point with a needle guard guide tube, without any therapeutic manoeuvre will be applied.
  Interventions: Procedure: Placebo Comparator: Placebo Gastrocnemius dry needling

INTERVENTIONS:
Procedure: Experimental: Deep dry needling — Deep dry needling until achieving twitch response of the muscle
  Arms: Deep dry needling
Procedure: Experimental: Superficial dry needling — Superficial dry needling to achieve sensitive pain with needle rotation
  Arms: Superficial dry needling
Procedure: Placebo Comparator: Placebo Gastrocnemius dry needling — Simulate pain with de plastic needle guard in the gastrocnemius muscle
  Arms: Placebo Gastrocnemius dry needling

SUMMARY:
This study investigates the effect of two different techniques (deep dry needling and superficial dry needling) on the latent myofascial trigger point in the upper trapezius. Subjects with latent Myofascial trigger point in this location of the muscle will be identified and will be randomly assigned to one out of the three groups: deep dry needling, superficial dry needling or sham dry needling in gastrocnemius muscle. cervical range of motion and pain pressure threshold in the upper trapezius will be registered before, immediately after the intervention, at 24 hours after the intervention, at 72 hours after the intervention and a week after the intervention

ELIGIBILITY:
Inclusion Criteria:

* Present the latent Myofascial trigger Point (MTP) 1 in upper trapezius.
* Accept participation in the study (signature of informed consent).
* Be in an age range between 18 and 55 years.
* Do not present any exclusion criteria.

Exclusion Criteria:

* Do not present MTP 1 latent in the upper trapezius.
* Suffering and / or having suffered from upper limb pathologies, deformities or orthopedic injuries that could alter the static and biomechanics of the shoulder and neck.
* Not clearly identify the MTP 1 in the upper trapezius.
* Have been diagnosed with fibromyalgia, myelopathy or radiculopathy.
* Having contraindicated the technique of dry needling for suffering, for example, coagulation problems.
* Having suffered a whiplash.
* Be pregnant.
* Have used analgesics 24 hours before participating in the study.
* Having belonephobia.
* Know the study techniques.
* Be in physiotherapy treatment and / or have been treated with needle techniques at some time.
* Having had cervical surgery.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2018-10-25 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | a week
  Amount of pressure (Kg/cm2) applied at the upper trapezius myofascial trigger point site that elicit pain for the patient will be reported

SECONDARY OUTCOMES:
Cervical range of motion | a week
  cervical movement in flexion and extension, left and right rotation and side bending left and right

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Montero-Navarro, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Universidad CEU Cardenal Herrera, Valencia, Moncada, Spain

REFERENCES:
- [Background] Segura-Orti E, Prades-Vergara S, Manzaneda-Pina L, Valero-Martinez R, Polo-Traverso JA. Trigger point dry needling versus strain-counterstrain technique for upper trapezius myofascial trigger points: a randomised controlled trial. Acupunct Med. 2016 Jun;34(3):171-7. doi: 10.1136/acupmed-2015-010868. Epub 2016 Jan 8. PMID 26746173
- [Background] Martin-Pintado-Zugasti A, Pecos-Martin D, Rodriguez-Fernandez AL, Alguacil-Diego IM, Portillo-Aceituno A, Gallego-Izquierdo T, Fernandez-Carnero J. Ischemic Compression After Dry Needling of a Latent Myofascial Trigger Point Reduces Postneedling Soreness Intensity and Duration. PM R. 2015 Oct;7(10):1026-1034. doi: 10.1016/j.pmrj.2015.03.021. Epub 2015 Mar 31. PMID 25836591
- [Background] Ziaeifar M, Arab AM, Karimi N, Nourbakhsh MR. The effect of dry needling on pain, pressure pain threshold and disability in patients with a myofascial trigger point in the upper trapezius muscle. J Bodyw Mov Ther. 2014 Apr;18(2):298-305. doi: 10.1016/j.jbmt.2013.11.004. Epub 2013 Nov 9. PMID 24725800
- [Background] Mejuto-Vazquez MJ, Salom-Moreno J, Ortega-Santiago R, Truyols-Dominguez S, Fernandez-de-Las-Penas C. Short-term changes in neck pain, widespread pressure pain sensitivity, and cervical range of motion after the application of trigger point dry needling in patients with acute mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Apr;44(4):252-60. doi: 10.2519/jospt.2014.5108. Epub 2014 Feb 25. PMID 24568260
- [Background] Llamas-Ramos R, Pecos-Martin D, Gallego-Izquierdo T, Llamas-Ramos I, Plaza-Manzano G, Ortega-Santiago R, Cleland J, Fernandez-de-Las-Penas C. Comparison of the short-term outcomes between trigger point dry needling and trigger point manual therapy for the management of chronic mechanical neck pain: a randomized clinical trial. J Orthop Sports Phys Ther. 2014 Nov;44(11):852-61. doi: 10.2519/jospt.2014.5229. Epub 2014 Sep 30. PMID 25269764
- [Result] Abbaszadeh-Amirdehi M, Ansari NN, Naghdi S, Olyaei G, Nourbakhsh MR. Therapeutic effects of dry needling in patients with upper trapezius myofascial trigger points. Acupunct Med. 2017 Apr;35(2):85-92. doi: 10.1136/acupmed-2016-011082. Epub 2016 Oct 3. PMID 27697768
- [Derived] Montero Navarro S, Del Rio Medina S, Martin Botella Rico J, Isabel Rocha Ortiz M, Teresa Perez Gracia M. Analysis and comparison of pain pressure threshold and active cervical range of motion after superficial and deep dry needling techniques of the upper trapezius muscle. Acupunct Med. 2022 Feb;40(1):13-23. doi: 10.1177/09645284211039523. Epub 2021 Sep 23. PMID 34553614
- See also: The University CEU-Cardenal Herrera is th first private university in the Valencian Community. It belongs to the Foundation San Pablo - CEU and is the leading educational organization in Spain with three Universities all over Spain — http://www.uchceu.es

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-12-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT03719352/Prot_SAP_ICF_000.pdf